CLINICAL TRIAL: NCT02577159
Title: Effects of Dapagliflozin on Hyperlipidemia, Glycemic Control and Insulin Resistance in Type 2 Diabetic Patients (DAPHNIS Study)
Brief Title: Dapagliflozin on Hyperlipidemia and Insulin Resistance in Type 2 Diabetic Patients (DAPHNIS Study)
Acronym: DAPHNIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osaka University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPHNIS
Record Dates: First submitted 2015-08-11; First posted 2015-10-16 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: sodium-glucose cotransporter 2 inhibitor; Diabetes Mellitus, Type 2; dyslipidemia; remnants; apolipoprotein B-48
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dapagliflozin (Experimental): Diabetic patients who met the inclusion/exclusion criteria. Dapagliflozin is orally administered for 8 weeks in the dose of 5mg per day if there is no serious event included in termination criteria. If the effect for improving diabetes is insufficient, it is allowed to raise its dose up to 10mg/day.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin is orally administered for 8 weeks in the dose of 5mg per day by adding the conventional treatment if there is no serious event included in termination criteria. If the effect for improving diabetes is insufficient, it is allowed to raise its dose up to 10mg/day.
  Other Names: conventional treatment

SUMMARY:
The investigators will investigate whether dapagliflozin (FORXIGA) might improve lipoprotein metabolism as well as hyperglycemia in Japanese patients with type II diabetes mellitus whose HbA1c levels are less than 7.0% (from 20 to 65 years of age). The investigators will examine changes of fasting lipoprotein profile including TG, TC, HDL-C, apoB-48 and RemL-C before and after the 8 weeks administration of dapagliflozin.

DETAILED DESCRIPTION:
In this study, the investigators will investigate whether dapagliflozin (FORXIGA) might improve lipoprotein metabolism as well as hyperglycemia in Japanese patients with type II diabetes mellitus. Primary Objective is to examine changes of fasting lipoprotein profile by the administration of dapagliflozin; Concentrations of apoB-48 and RemL-C. Secondary Objectives are; to examine changes of fasting glucose and HbA1c (NGSP) level by the administration of dapagliflozin, to examine changes of fasting lipid profile by the administration of dapagliflozin; Concentrations of TG, TC, HDL-C and LDL-C, to examine changes of fractions of free fatty acids, protein mass of LPL, and lipoprotein profile assessed by the HPLC by the administration of dapagliflozin, to examine changes of biomarkers for renal and hepatic function by the administration of dapagliflozin, and to examine the frequency of adverse effects by the administration of dapagliflozin. This study is open-label study and contains patients who are diabetes mellitus of from 20 to 65 years of age and their Patients who have not achieve the clinical target of the glycemic control (less than 7.0% in HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with type 2 diabetes mellitus of from 20 to 65 years of age.
* Patients who have not achieve the clinical target of the glycemic control (less than 7.0% in HbA1c).
* Patients who received the diet therapy, the exercise therapy or the following anti-diabetic drugs in addition to the diet and/or exercise therapy (up to two drugs) with dosage stable for 8 weeks prior to entry.
* Sulfonylurea (Glymepiride 2mg/day or less, Glibenclamide 1.25mg/day or less, Gliclazide 40mg/day or less)
* Thiazolidine (Actos)
* Biguanide (Metformin, Buformin)
* alpha-glucosidase inhibitor (Voglibose, Miglitol, Acarbose)
* DPP4 inhibitors (Sitagliptin, Linagliptin, Anagliptin, Teneligliptin, Alogliptin, Saxagliptin)
* Informed consent to participate in the study prior to any study procedures.

Exclusion Criteria:

* Type 1 diabetes mellitus
* Moderate or severe renal dysfunction (eGFR<45 ml/min/1.73m2 or hemodialysis)
* Severe hepatic insufficiency (AST and/or ALT >3x upper limit of normal)
* Adrenal insufficiency or pituitary gland dysfunction
* Malnourishment, starvation, irregular dietary intake, poor dietary intake, debilitating condition or a severe muscle movement
* Volume depleted patients; concomitant medication such as loop diuretics.
* Excessive alcohol intake (>60g daily)
* SGLT2 inhibitors such as dapagliflozin are already administered
* Contraindication with dapagliflozin
* Start a new medication of statins, fibrates, ezetimibe or probucol within a month
* Females who are likely to be pregnant, during pregnancy or lactating
* Participants in other clinical trials
* Inability to communicate and comply with all study requirements.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07-01; Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in fasting lipoprotein profiles | at four and eight weeks after the administration of dapagliflozin
  Changes in fasting lipoprotein profiles including concentrations of apoA-1, apoA-2, apoB, apoB-48, apoC-2, apoC-3, apoE, RemL-C, free-fatty acids profile, LPL protein mass and lipoprotein profile assessed by the HPLC at four and eight weeks after the administration of dapagliflozin

SECONDARY OUTCOMES:
Changes in fasting lipid profiles | at four and eight weeks after the administration of dapagliflozin
  Changes in fasting lipid profiles including concentrations of triglyceride(TG), total cholesterol(TC), HDL-cholesterol (HDL-C) and LDL-C at four and eight weeks after the administration of dapagliflozin
Changes in fasting blood glucose and HbA1c | at four and eight weeks after the administration of dapagliflozin
  Changes in fasting blood glucose and HbA1c at four and eight weeks after the administration of dapagliflozin
Changes in insulin and adiponectin | at four and eight weeks after the administration of dapagliflozin
  Changes in other clinical profiles including concentrations of insulin and adiponectin
Frequency of adverse side effects | at four and eight weeks after the administration of dapagliflozin
  Frequency of adverse side effects at four and eight weeks after the administration of dapagliflozin
Changes in biomarkers for renal and hepatic function | four and eight weeks after the administration of dapagliflozin.
  Changes in biomarkers for renal and hepatic function at four and eight weeks after the administration of dapagliflozin.

CONTACTS AND LOCATIONS:
Overall Officials: Shizuya Yamashita, MD, PhD, Principal Investigator — Osaka University Graduate School of Medicine
Locations (3):
- Japan (3):
  - Sousei Hospital, Kadoma, Osaka
  - Osaka Central Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka

REFERENCES:
- [Background] Hanada H, Mugii S, Okubo M, Maeda I, Kuwayama K, Hidaka Y, Kitazume-Taneike R, Yamashita T, Kawase R, Nakaoka H, Inagaki M, Yuasa-Kawase M, Nakatani K, Tsubakio-Yamamoto K, Masuda D, Ohama T, Matsuyama A, Ishigami M, Nishida M, Komuro I, Yamashita S. Establishment of chemiluminescence enzyme immunoassay for apolipoprotein B-48 and its clinical applications for evaluation of impaired chylomicron remnant metabolism. Clin Chim Acta. 2012 Jan 18;413(1-2):160-5. doi: 10.1016/j.cca.2011.09.013. Epub 2011 Sep 19. PMID 21958700
- [Background] Masuda D, Sakai N, Sugimoto T, Kitazume-Taneike R, Yamashita T, Kawase R, Nakaoka H, Inagaki M, Nakatani K, Yuasa-Kawase M, Tsubakio-Yamamoto K, Ohama T, Nakagawa-Toyama Y, Nishida M, Ishigami M, Masuda Y, Matsuyama A, Komuro I, Yamashita S. Fasting serum apolipoprotein B-48 can be a marker of postprandial hyperlipidemia. J Atheroscler Thromb. 2011;18(12):1062-70. doi: 10.5551/jat.10470. Epub 2011 Sep 24. PMID 21946533
- [Background] Okubo M, Hanada H, Matsui M, Hidaka Y, Masuda D, Sakata Y, Yamashita S. Serum apolipoprotein B-48 concentration is associated with a reduced estimated glomerular filtration rate and increased proteinuria. J Atheroscler Thromb. 2014;21(9):974-82. doi: 10.5551/jat.23309. Epub 2014 Jun 2. PMID 24882621
- [Background] Mugii S, Hanada H, Okubo M, Masuda D, Takeoka K, Hidaka Y, Ohama T, Matsuyama A, Nakagawa-Toyama Y, Nishida M, Ishigami M, Komuro I, Yamashita S. Thyroid function influences serum apolipoprotein B-48 levels in patients with thyroid disease. J Atheroscler Thromb. 2012;19(10):890-6. doi: 10.5551/jat.12757. Epub 2012 Jul 4. PMID 22786447
- [Background] Nakatani K, Sugimoto T, Masuda D, Okano R, Oya T, Monden Y, Yamashita T, Kawase R, Nakaoka H, Inagaki M, Yuasa-Kawase M, Tsubakio-Yamamoto K, Ohama T, Nishida M, Ishigami M, Komuro I, Yamashita S. Serum apolipoprotein B-48 levels are correlated with carotid intima-media thickness in subjects with normal serum triglyceride levels. Atherosclerosis. 2011 Sep;218(1):226-32. doi: 10.1016/j.atherosclerosis.2011.05.009. Epub 2011 May 18. PMID 21641598
- [Background] Masuda D, Sugimoto T, Tsujii K, Inagaki M, Nakatani K, Yuasa-Kawase M, Tsubakio-Yamamoto K, Ohama T, Nishida M, Ishigami M, Kawamoto T, Matsuyama A, Sakai N, Komuro I, Yamashita S. Correlation of fasting serum apolipoprotein B-48 with coronary artery disease prevalence. Eur J Clin Invest. 2012 Sep;42(9):992-9. doi: 10.1111/j.1365-2362.2012.02687.x. Epub 2012 May 15. PMID 22587365
- [Background] Ji L, Ma J, Li H, Mansfield TA, T'joen CL, Iqbal N, Ptaszynska A, List JF. Dapagliflozin as monotherapy in drug-naive Asian patients with type 2 diabetes mellitus: a randomized, blinded, prospective phase III study. Clin Ther. 2014 Jan 1;36(1):84-100.e9. doi: 10.1016/j.clinthera.2013.11.002. Epub 2013 Dec 28. PMID 24378206
- [Background] Kaku K, Maegawa H, Tanizawa Y, Kiyosue A, Ide Y, Tokudome T, Hoshino Y, Yang J, Langkilde AM. Dapagliflozin as monotherapy or combination therapy in Japanese patients with type 2 diabetes: an open-label study. Diabetes Ther. 2014 Dec;5(2):415-33. doi: 10.1007/s13300-014-0086-7. Epub 2014 Oct 24. PMID 25341477
- [Background] Bolinder J, Ljunggren O, Kullberg J, Johansson L, Wilding J, Langkilde AM, Sugg J, Parikh S. Effects of dapagliflozin on body weight, total fat mass, and regional adipose tissue distribution in patients with type 2 diabetes mellitus with inadequate glycemic control on metformin. J Clin Endocrinol Metab. 2012 Mar;97(3):1020-31. doi: 10.1210/jc.2011-2260. Epub 2012 Jan 11. PMID 22238392